CLINICAL TRIAL: NCT05742256
Title: Effect of Oxycodone Combined With Ultrasound Guided Thoracic Paravertebral Nerve Block on Postoperative Analgesia in Patients With Lung Cancer Undergoing Thoracoscopic Surgery
Brief Title: Oxycodone in Combination With Parathoracic Nerve Block is Used for Postoperative Analgesia in Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Pengcai Shi, Chief physician，Master Tutor, Qianfoshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YXLL-KY-2022(116)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Oxycodone
Keywords: Oxycodone; Postoperative analgesia; lung cancer; thoracic paravertebral nerve block
MeSH Terms: conditions — Lung Neoplasms | interventions — Oxycodone; Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test group 1(OCA group) (Experimental)
  Interventions: Drug: Oxycodone 1mg/kg
- Test group 2(OCB group) (Experimental)
  Interventions: Drug: Oxycodone 1.5mg/kg
- Control group(SF group) (Active Comparator)
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Oxycodone 1mg/kg — Test group 1 (OCA group):oxycodone 1mg/kg + flurbiprofen 50mg + ondansetron 16mg + 0.9% normal saline diluted to 100ml
  Other Names: Oxycodone
  Arms: Test group 1(OCA group)
Drug: Oxycodone 1.5mg/kg — Test group 2 (OCB group): oxycodone 1.5mg/kg + flurbiprofen 50mg + ondansetron 16mg + 0.9% normal saline diluted to 100ml.
  Arms: Test group 2(OCB group)
Drug: Sufentanil — Control group (SF group): sufentanil 2ug/kg + flurbiprofen + ondansetron 16mg + 0.9% normal saline diluted to 100ml.
  Arms: Control group(SF group)

SUMMARY:
In this study, the effect of oxycodone combined with ultrasound-guided paravertebral nerve block on the postoperative analgesic effect of thoracoscopic lung cancer was investigated, and the effect and reasonable dose of oxycodone were explored, which provided a reference for the clinical multimodal analgesia after thoracoscopic lung cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age > 60 years
2. Patients undergoing thoracoscopic lobectomy
3. ASA (American Academy of Anesthesiologists) Grades I-III
4. There were no obvious abnormalities in heart, liver, and kidney function
5. Sign the informed consent form for this clinical study

Exclusion Criteria:

1. History of oxycodone or sufentanil allergy
2. Renal or hepatic dysfunction
3. History of drug or alcohol abuse
4. Psychiatric disorders: schizophrenia, epilepsy, Parkinson's disease, myasthenia gravis
5. Those who have difficulty communicating due to coma, severe dementia, speech barrier, or those who cannot cooperate due to other diseases.
6. People with head trauma or other brain diseases -

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The main indicators were NRS scores at rest and cough at 24 h postoperatively. | at 24h after surgery
  NRS (numerical rating scale) is composed of 11 numbers from 0 to 10, and patients use 11 numbers from 0 to 10 to describe the intensity of pain, and the higher the number, the more severe the pain.

SECONDARY OUTCOMES:
Time to double-lumen tracheal extraction | Within two hours after surgery
  Time to double-lumen tracheal extraction
NRS score at rest and cough | at 2h , 4h, 12h, 48h after surgery
  NRS (numerical rating scale) is composed of 11 numbers from 0 to 10, and patients use 11 numbers from 0 to 10 to describe the intensity of pain, and the higher the number, the more severe the pain.
sedation score (Ramsay sedation score) | at 2 h , 4 h , 12 h ,24 h,48 h postoperatively
  The Ramsay sedation score is the most widely used sedation scoring criterion in clinical practice. It is divided into six levels, reflecting three levels of wakefulness and three levels of sleep. The higher the level, the deeper the level of sedation.
sufentanil consumption | Within 48 hours after surgery
  sufentanil consumption
oxycodone consumption | Within 48 hours after surgery
  oxycodone consumption
analgesic pump compressions | Within 48 hours after surgery
  analgesic pump compressions
additional analgesic doses | Within 48 hours after surgery
  additional analgesic doses
incidence of adverse reactions: nausea, vomiting, respiratory depression, dizziness, itchin | Within 48 hours after surgery
  incidence of adverse reactions: nausea, vomiting, respiratory depression, dizziness, itchin
gastrointestinal recovery (exhaust time) | Within 48 hours after surgery
  gastrointestinal recovery (exhaust time)
laboratory results of C-reactive protein 1 day before and after surgery | Within 48 hours after surgery
  laboratory results of C-reactive protein 1 day before and after surgery
laboratory results of interleukin-6 laboratory test 1 day before and after surgery | Within 48 hours after surgery
  laboratory results of interleukin-6 laboratory test 1 day before and after surgery

REFERENCES:
- [Derived] Wang Y, Wu G, Liu Z, Wei X, Feng H, Su J, Shi P. Effect of oxycodone combined with ultrasound-guided thoracic paravertebral nerve block on postoperative analgesia in patients with lung cancer undergoing thoracoscopic surgery: protocol for a randomised controlled study. BMJ Open. 2023 Oct 16;13(10):e074416. doi: 10.1136/bmjopen-2023-074416. PMID 37844986